CLINICAL TRIAL: NCT05231928
Title: Efficacy of a Novel Argon Laser Iridoplasty for Management of Pigment Dispersion Syndrome Assessed by Anterior Segment Optical Coherence Tomography
Brief Title: A Novel Argon Laser Iridoplasty for Pigment Dispersion Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Mohamed Ameen Ismail, Research assistant of ophthalmology, Fayoum University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R 211
Record Dates: First submitted 2022-01-30; First posted 2022-02-09 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Pigment Dispersion Syndrome; Pigmentary Glaucoma
MeSH Terms: conditions — Glaucoma-Related Pigment Dispersion Syndrome; Glaucoma, Open-Angle

STUDY DESIGN:
Intervention Model Description: Interventional, longitudinal, prospective, uncontrolled case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Argon Laser Iridoplasty (Experimental): Argon Laser is applied to the anterior iris surface after pharmacological miosis and instillation of ocular surface anesthetic using YAG capsulotomy lens or Abraham Iridotomy lens as auxiliary lenses. Laser is applied at sites and with parameters that are tailored for each case according to exact iris configuration, iris colour and pupil diameter.
  Interventions: Procedure: Argon Laser Iridoplasty

INTERVENTIONS:
Procedure: Argon Laser Iridoplasty — Argon Laser is applied to the anterior iris surface at sites and with parameters tailored according to iris configuration, pupil size, iris colour.
  The device used is Nidek Argon Laser device with YAG capsulotomy or Abraham Iridotomy lens as auxilliary lenses.
  -Topical Pilocarpine 2% and ocular surface anesthetic are applied prior to the procedure and Brimonidine 0.2% bid is used fo a week after the procedure together with topical dexamethasone ophthalmic solution.

SUMMARY:
Pigment dispersion syndrome is a rare condition where anomalous iris configuration leads to posterior iris bowing with subsequent friction with the lenticulozonular unit resulting in dispersion of pigment from the back surface of the iris into the anterior segment as well as thinning with resultant transillumination defects in the mid iris segment. The released pigment is deposited in various parts of the anterior segment resulting in a constellation of clinical signs:

Krukenberg Spindle: Back surface of the cornea Zentmayer ring: Back surface of the lens. Egger line: Anterior vitreous face. More importantly, pigment accumulated in the trabecular meshwork leading to visible hyperpigmentation of the trabeculum seen by gonioscopy. This leads to reduction of aqueous outflow which leads to ocular hypertension or even glaucoma which is known as pigment dispersion glaucoma which is considered one of refractory glaucomas.

Current practice in the management of pigment dispersion syndrome revolves around the management of glaucoma when it develops by IOP lowering medication, Laser trabeculoplasty or peripheral iridoplastyor glaucoma surgery as a last resort. The only prophylactic measure in practice that is aimed at preventing the progression from mere pigment dispersion to pigment dispersion glaucoma is the long term use of miotic eyedrops e.g. Pilocarpine which comes with both risks and side effects i.e. the risk of retinal breaks and detachment which is even higher in a cohort which is predominantly myope, the constriction of visual field and ocular surface complications.

In this interventional case series, the investigators assess the efficacy of a novel Argon Laser iridoplasty in the management of pigment dispersion through correcting the posterior iris bowing and hence halting the dispersion process so that glaucoma wouldn't develop in the first place instead of managing glaucoma after it sets in which proved refractory.

DETAILED DESCRIPTION:
*Study design: Interventional, longitudinal, prospective, uncontrolled case series study

**Methods:

* Population: cases of pigment dispersion syndrome/glaucoma.
* Sample size:

Not determined since it is a case series with still active recruitment.

* A series of pigment dispersion syndrome and/or pigment dispersion glaucoma cases encountered in the ophthalmology outpatient clinic of Fayoum University Hospitals will be assessed clinically for confirmation of signs of pigment dispersion by slitlamp examination and gonioscopy. Intraocular pressure will be measured and monitored. Fundus examination with special attention to the optic disc will be done. Cases will be assessed prior to iridoplasty by anterior segment optical coherence tomography to document the anomalous iris configuration with subsequent serial anterior segment OCT at one week, one month and three months after iridoplasty as well as IOP measurement.
* The iridoplasty procedure will be performed as follows:

  1. Pilocarpine 2% topically is used to induce miosis.
  2. Topical ocular anesthetic is instilled.
  3. The Nidek Argon laser device together with a YAG capsolutomy or Abraham Iridotomy lens as auxilliary lenses are used.
  4. The site and parameters of argon laser applications on the anterior iris surface are tailored for each patient according to iris configuration and pupil diameter in mesopic conditions determined by anterior segment OCT.
  5. Topical Brimonidine 0.2% bid is used for one week after the procedure to guard against IOP spikes.

ELIGIBILITY:
Inclusion Criteria:

* Pigment dispersion syndrome/glaucoma confirmed by either clinical signs or imaging with documented posterior iris bowing.

Exclusion Criteria:

* Active or history of Uveitis.
* Pupil size > 7mm in mesopic conditions.
* Previous Iris-based laser procedures e.g. Iridotomy, Iridoplasty

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
correction of posterior iris bowing | Baseline documentation of posterior bowing by anterior segment OCT followed by one week, one month, three months follow up by anterior segment OCT for changes in iris configuration.
  The posterior iris bowing is at the basis of pigment dispersion pathology and so the correction of this posterior bowing halts the disease process at its very roots.
  Correction means either flattening or anterior bowing of iris (a change from negative bowing values to zero bowing or positive bowing values)

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University Hospitals, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No